CLINICAL TRIAL: NCT04540588
Title: A Safety and Efficacy Study of Retreatment With Intratumoral Diffusing Alpha Radiation Emitters
Brief Title: Retreatment With Intratumoral Diffusing Alpha Radiation Emitters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-CMN-05
Record Dates: First submitted 2020-08-18; First posted 2020-09-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Skin Cancer; Mucosal Neoplasm of Oral Cavity; Soft Tissue Neoplasm
Keywords: Squamous Cell Carcinoma; SCC; Skin Cancer; Skin metastasis; HNSCC; Carcinoma, Squamous; CMN; Basal cell carcinoma; Superficial sarcoma; Kaposi sarcoma; Alpha radiation; Cutaneous lesion; Tongue cancer; Lip cancer; Brachytherapy; Recurrent disease; Persistent lesion
MeSH Terms: conditions — Skin Neoplasms; Soft Tissue Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Basal Cell; Sarcoma, Kaposi; Tongue Neoplasms; Lip Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.
  Other Names: DaRT

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for superficial cutaneous, mucosal or soft tissue neoplasia

DETAILED DESCRIPTION:
This will be a prospective, open label, single arm, controlled study, assessing the safety and efficacy of re-treatment with diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive seeds inserted into the tumor.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Superficial lesions with histopathological confirmation of either recurrent or persistent disease following DaRT treatment. .

Reduction in tumor size 70 days after DaRT insertion will be assessed. Safety will be assessed by the incidence, severity and frequency of all Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathological confirmation of either recurrent or persistent disease following DaRT treatment.
* Subjects with a tumor size ≤ 5 centimeters in the longest diameter.
* Target lesion technically amenable for full coverage with the Alpha DaRT seeds.
* Brachytherapy indication validated by a multidisciplinary team.
* Measurable disease according to RECIST v1.1.
* Subjects over 18 years old.
* Subjects' ECOG Performance Status Scale is < 2.
* Subjects' life expectancy is more than 6 months.
* Platelet count ≥100,000/mm3.
* AST and ALT ≤ 2.5 X ULN
* WBC ≥ 3500/μl, granulocyte ≥ 1500/μl
* International normalized ratio of prothrombin time ≤1.4 for patients not on Warfarin
* Creatinine ≤2.3 mg/dL.
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test before the Ra-224 implantation and are required to use an acceptable contraceptive method to prevent pregnancy for 3 months after brachytherapy.
* Subjects are willing to sign an informed consent form.

Exclusion Criteria:

* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids
* Known hypersensitivity to any of the components of the treatment.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT
* High probability of protocol non-compliance (in opinion of investigator)
* Subjects not willing to sign an informed consent
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Tumor response to DaRT | 9-11 weeks post DaRT insertion
  Assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)
Adverse events | From conscent up to 9-11 weeks post DaRT insertion
  Frequency, severity and causality of acute adverse events related to the DaRT treatment. Adverse events will be assessed and graded according to Common Terminology and Criteria for adverse events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Change in tumor volume | 9-11 weeks post DaRT insertion
  Based on imaging
Local control rate | 9-11 weeks post DaRT insertion
  Will be assessed as the number of complete responses, partial responses and stable disease divided by the total numbers of tumors treated.

OTHER OUTCOMES:
Adverse Events | From conscent up to 9-11 weeks post DaRT insertion
  Incidence of all Adverse Events (AE) related and unrelated to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aron Popovtzer, M.D, Principal Investigator — Sharett institute, Hadassah Medical Center - Ein-Kerem
Locations (1):
- Sharett institute, Hadassah University Hospital - Ein-Kerem, Jerusalem, Israel